CLINICAL TRIAL: NCT02390869
Title: A Randomized Phase III Multicenter Trial Assessing Efficacy and Toxicity of a Combination of Rituximab and Lenalidomide (R2) vs Rituximab Alone as Maintenance After Chemoimmunotherapy With Rituximab-chemotherapy (R-CHT) for Relapsed/Refractory FL Patients Not Eligible for Autologous Transplantation (ASCT).
Brief Title: Rituximab and Lenalidomide vs Rituximab Alone as Maintenance After R-chemoterapy for Relapsed/Refractory FL Patients
Acronym: FIL_RENOIR12
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIL_RENOIR12
Record Dates: First submitted 2015-03-02; First posted 2015-03-18 (Estimated); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Lymphoma, Follicular
Keywords: relapse/refractory
MeSH Terms: conditions — Lymphoma, Follicular; Recurrence | interventions — Rituximab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- R2-MANT (Experimental): A) Rituximab B) Lenalidomide
  Interventions: Drug: R2-MANT
- R-MANT (Active Comparator): A) Rituximab
  Interventions: Drug: R-MANT

INTERVENTIONS:
Drug: R2-MANT — A) Rituximab 375 mg/sqm on day 1 every 90 days for 8 cycles B) Lenalidomide (10 mg daily on days 1-21 every 28 days) for 24 cycles
  Other Names: Rituximab and Lenalidomide (R2)
  Arms: R2-MANT
Drug: R-MANT — A) Rituximab 375 mg/sqm on day 1 every 90 days for 8 cycles
  Other Names: Rituximab (R)
  Arms: R-MANT

SUMMARY:
A randomized phase III multicenter trial assessing efficacy and toxicity of a combination of Rituximab and Lenalidomide (R2) vs Rituximab alone as maintenance after chemoimmunotherapy with Rituximab-chemotherapy (R-CHT) for relapsed/refractory FL patients not eligible for autologous transplantation (ASCT)

DETAILED DESCRIPTION:
Among Non-Hodgkin lymphomas (NHL), Follicular Lymphoma (FL) is the second one in terms of frequency, accounting for about 25% of all NHL cases in the western hemisphere. A predominance in females is reported, and the median age at the diagnosis is 60 years.

FL cells originates from normal counterparts germinal B cells. At a molecular level, the pathology is thought to be dependent on multiple DNA alterations. However, a large amount of patients (approximately 85%) have t(14;18), with a consequent overexpression of anti-apoptotic protein BCL-2.

An additional hallmark of pathology is bone marrow involvement (70% of patients), while this is seldom noticed in other organs. Finally, 20% of patients show high levels of serum lactate dehydrogenase (LDH) and/or B symptoms.

FL is actually considered an incurable disease. Although FL responds well to initial chemotherapy, most patients will eventually relapse, requiring multiple subsequent therapeutic regimens during the course of disease to achieve new period of remission, that are nevertheless shorter. Relapsed/refractory FL in advanced stage, especially in older patients, has a relatively poor prognosis, and several patients die for infectious complications and/or progressive disease. This subset of patients usually do not survive more than 5 years.

Thus there is a need for new, less toxic and more active treatment in particular for patients with recurrent disease. The addition of Rituximab to chemotherapy showed a clear benefit in terms of overall response rate, quality of response, event-free survival and, in most studies, overall survival; nevertheless, relapses still occur. Moreover Rituximab also proved highly effective when employed as maintenance treatment either following chemotherapy or Rituximab-supplemented chemotherapy. The success of Rituximab maintenance led to the widespread opinion that in the context of indolent lymphomas novel "smart" drugs characterized by a good safety profile need to be carefully evaluated not only in the induction but also in the maintenance setting.

Autologous stem cell transplantation and radioimmunotherapy are therapeutic option for relapsed/refractory FL patients, but can be considered only for younger or fit patients and can be delivered only in large institutions.

Therefore the search of new, more manageable, therapeutic agents with different mechanisms of action, especially for elderly or frail patients, is ongoing.

Bendamustine is highly effective in relapsed/refractory indolent non-Hodgkin lymphoma (NHL) and Mantle Cell Lymphoma (MCL), including patients who are refractory to rituximab and those previously treated with other alkylating agents. Therefore, bendamustine is now widely used in this setting and provides another effective treatment option for patients who progress after CHOP-R. Two phase II studies have combined bendamustine (90 mg/m2 days 2-3 every 28 days) with rituximab (375 mg/m2 day 1) and both reported similar results. The overall response rate was 90% (60% CR) for the entire patient population, and median Progression-free survival (PFS) for all patients was 24 months. Based on these encouraging results in the relapsed/refractory setting, the Study group indolent Lymphomas (StiL) initiated a large, randomized, phase III trials of bendamustine (90 mg/m2 days 1-2 every 28 days) plus rituximab (375 mg/m2 day 1). This trial compared B-R with standard CHOP-R (21-day cycles) in previously untreated patients with indolent NHL and MCL. 549 patients with predominantly stage IV disease were enrolled, and the treatment groups were well balanced for all baseline characteristics. Approximately 55% of patients had FL, approximately 20% had MCL, and the remaining 25% had other indolent lymphomas. Although the overall response rate was similar in the B-R and CHOP-R arms (93.8% and 93.5%, respectively), the CR rate was significantly higher in the B-R arm (40.1% compared with 30.8% for CHOP-R; P .03), and the median PFS was significantly longer in the B-R arm (54.8 months v 34.8 months for CHOP-R; P .0002). No difference in survival has been observed thus far, further follow-up of this ongoing study will be required to address whether B-R improves survival compared with CHOP-R. Nevertheless, bendamustine plus rituximab yielded more durable responses and improved PFS compared with CHOP-R in previously untreated patients with indolent lymphomas. Moreover, bendamustine plus rituximab was better tolerated.

Lenalidomide is an immunomodulatory agent with multiple mechanisms of action wich include antiproliferative activity as well as microenvironmental effects such as inhibition angiogenesis and stimulation of T-cell mediated response. Lenalidomide given as monotherapy proved to be active, with an acceptable toxicity profile, in B-cell malignancies such as multiple myeloma, chronic lymphocytic leukemia, mantle cell lymphoma and diffuse large B-cell lymphoma.

Recent reports on Lenalidomide in FL, both for untreated and relapsed patients, are promising.

Forty-three patients with relapsed or refractory indolent non Hodgkin's lymphoma (NHL) were treated with oral Lenalidomide 25 mg once daily on days 1 to 21 of every 28-day cycle for 52 weeks or until progression. Twenty-two of the 43 patients enrolled had FL In this subgroup overall response rate was 27%, with a 9% complete remission rate. Most common adverse events were myelosuppression, fatigue, gastrointestinal events and cutaneous rash, while predominant grade 3/4 serious adverse events were neutropenia and thrombocytopenia. Despite a median duration of response longer than 16.5 months, there was a disappointing median progression-free survival of 4.4 months.

Witzig et al. focused on Lenalidomide 25 mg in monotherapy in relapsed/refractory B-cell lymphomas. The cohort of patients was 217, 19 of them had a stage III FL. Regarding this patients subset, ORR was 42%, CR/Cru was 11%, median PFS was 8.9 months, median duration of response was not reached.

The cytotoxic effect of Rituximab appears to involve CDC, ADCC and induction of apoptosis. Early studies of Lenalidomide show the potential for high CR rates and long duration of response in FL and Chronic lymphocytic leukemia (CLL). Recent data suggest that the modulation of effector cells by Lenalidomide can enhance the antitumor activity of Rituximab and partially overcome its resistance in cell lines of relapsed/refractory NHL. Lenalidomide appears in fact to greatly enhance the monocyte and NK-mediated ADCC exerted by Rituximab, resulting in an increase of cancer cell killing compared to the single drugs. A synergistic activity between Rituximab and Lenalidomide has been reported in vitro in lymphoma cells and in animal models. Rituximab-lenalidomide (R2) combination has been consequently tested in clinical trials, including untreated or relapsed/refractory indolent NHL, with encouraging results.

The first report about the R2 combination in FL was presented at the 51th ASH meeting by Dutia M et al. Sixteen patients with relapsed/refractory indolent NHL have been treated with R2 combination, obtaining a 75% overall response (ORR) rate with an acceptable toxicity; interestingly, efficacy data seem better in FL patients with a 88% ORR. Moreover, in the unfavourable subgroups of rituximab refractory and heavily pre-treated patients, ORR rates were 57% and 70%, respectively. Estimated progression-free survival for all patients is 12 months. The major limitation of the study was the small number of patients, with only 9 FL patient included in the study.

Twenty-four patients with indolent B-cell lymphoma, previously resistant to Rituximab, received a Rituximab-Lenalidomide +/- Dexamethasone combination until progression of disease or unacceptable toxicity; Lenalidomide was administered at the dosage of 10 mg, 28 days per course. 28 over 45 patients had FL. No further FL group analysis were reported, but the study allowed to assess that also patients resistant to Rituximab in mono-therapy can benefit from R2, with or without Dexamethasone, achieving higher ORR (~61%) with relatively durable responses.

One hundred patients with stage III-IV untreated indolent NHL received the R2 combination in cycles of 28 days (Lenalidomide 20 mg orally once a day from day 1 to day 21 and Rituximab 375 mg/m2 intravenously on day 1). 49 patients (49%) composed the FL subset.

The outcome of FL patients was extremely positive, considering the ORR (98%) and the CR/CRu (85%). Moreover, when the R2 treatment was prolonged after 6 courses, a significant improvement was seen for CR/CRu. Finally, the PFS was 83% for FL patients after 24 months, and the toxicity profile was acceptable.

In CALGB 50401 randomized study 89 recurrent FL patients were treated with Lenalidomide alone versus R2 combination. ORR were 49% vs 75% and EFS was 1.2 vs 2.0 with a median follow up of 1.5 years.

Basing on these promising data, other trials proposed the combination of Lenalidomide and R-CHOP (R2-CHOP), as R-CHOP is the standard treatment for most patients with B-cell lymphomas. Briefly, both Phase I and Phase I/II trials confirmed the potential of the novel combination, although a large multi-centre trial is required to confirm the results.

ELIGIBILITY:
Inclusion Criteria:

* Follicular lymphoma grade I, II and IIIa according to the WHO classification. Rebiopsy at study entry is strongly encouraged but mandatory only in case of suspected transformation (elevated LDH or rapidly-growing disease or unusual relapse presentation).
* First or second relapse or progression following R-chemotherapy (Rituximab maintenance and IF radiotherapy are not considered treatment lines).
* Previous treatment with Bendamustine can be considered eligible if relapse occurred after ≥ 24 months.
* Age >18 years.
* Patients not eligible for high dose chemotherapy and ASCT because of: age ≥ 65 years, impaired PS or organ function due to major comorbidities or relapsed or refractory disease after previous ASCT before 65 of age.
* Stage II, III or IV according to Ann Arbor at relapse.
* Need of treatment according to SIE-SIES-GITMO guidelines for follicular lymphoma: stage II-IV with systemic symptoms, high tumor burden (i.e. >3 lymph nodes measuring >3 cm or a single lymph node >7 cm), extranodal disease, cytopenia due to marrow involvement, spleen involvement (≥16 cm by CT), leukemic phase, serious effusion, symptomatic or life endangering organ involvement, rapid lymphoma progression, consistently increased LDH levels.
* Must be able to adhere to the study visit schedule and other protocol standards.
* ECOG performance status ≤ 2 (except when PS impairment is related to lymphoma).
* Be willing and able to comply with the protocol for the duration of the study.
* Absolute neutrophil count (ANC) ≥ 1.5 x 10 9/L unless due to marrow involvement by lymphoma; and platelets count ≥ 75 x 109/L unless due to marrow involvement by lymphoma.
* Calculated creatinine clearances ≥ 40 ml/min.
* Agree to be using effective contraception for the entire treatment period according to standard guidelines for patients receiving lenalidomide

Exclusion Criteria:

* Any lymphoma subtype other than FL including transformed FL
* Grade 3b follicular lymphoma.
* Radiotherapy within 3 months prior to study entry
* Major surgery (excluding lymph node biopsy) within 28 days prior to registration.
* HIV positive serology. HBV and HCV positive patients will be not excluded from the study if the hepatic enzymes are within the ranges later defined. HBV occult carriers patients will be given lamivudine as prophylaxis starting one week before chemotherapy. HbsAg, HBcAb, HBV-DNA and HCV-RNA levels will be monitored twice every month in HCV or HBV positive patients.
* Life expectancy < 6 months.
* Known sensitivity or allergy to murine products.
* Prior history of malignancies, other than follicular lymphoma, unless the subject has been free of the disease for > 3 years with the exception of adequately cured localized non-melanoma skin cancer, carcinoma in situ of the cervix, carcinoma in situ of the breast or incidental histological finding of prostate cancer (TNM stage of T1a or T1b)
* Prior use of lenalidomide.
* Neuropathy > Grade 1.
* Myocardial infarction within the last 6 months
* Presence or history of CNS involvement by lymphoma.
* Subjects who are at a high risk for a thromboembolic event and are not willing to take venous thromboembolic (VTE) prophylaxis.
* Serum aspartate transaminase (AST/SGOT) or alanine transaminase (ALT/SGPT) > 3x upper limit of normal (ULN), except in subjects with documented liver involvement by lymphoma
* Total bilirubin > 2.0 mg/dl (34 umol/L) except in cases of Gilberts Syndrome and documented liver involvement by lymphoma
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Pregnant or lactating females.
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study, or which confounds the ability to interpret data from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
PFS | 2 years from randomization
  Progression-free survival

SECONDARY OUTCOMES:
OS | 2 years from randomization
  Overall survival
Toxicity (Common Terminology Criteria for Adverse Event version 4.03 (CTCAE) | 2 years from randomization
  classified according to definitions of Common Terminology Criteria for Adverse Event version 4.03 (CTCAE). It will be determined by the incidence of severe, life- threatening (CTCAE grade 3, 4 and 5) and/or serious adverse events (Infusion-related reactions).
Rate of molecular remission | 2 years from randomization
  proportion of patients PCR negative for Bcl-2/IgH at different time-points including those achieving continuous MR in two or more consecutive time-points
Rate of molecular conversion | 2 years from randomization
  proportion of patients from baseline PCR-positivity to PCR-negativity.
Rate of molecular relapse | 2 years from randomization
  proportion of patients from PCR-negativity to PCR-positivity.
Quality of Life(QoL) | 2 years from randomization
  using the EORTC QLQ-C30C questionnaire
The incremental cost-effectiveness ratio | 2 years from randomization
  Quality Adjusted Life Years (QALYs) using Euro-Qol (EQ-5D) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Umberto Vitolo, MD, Study Chair — Candiolo Cancer Institute, FPO-IRCCS
Locations (28):
- Italy (28):
  - ASST Grande Ospedale Metropolitano Niguarda, Milan, MI
  - AUSL di Ravenna, Ravenna, RA
  - Fondazione Del Piemonte Per L'Oncologia Ircc Di Candiolo, Candiolo, Torino
  - Ospedale S. Giacomo di Castelfranco Veneto, Castelfranco Veneto, Treviso
  - A.O. S. Maria di Terni, Terni, TR
  - ASST Valle Olona - Ospedale di Circolo di Busto Arsizio, Busto Arsizio, Varese
  - Ospedale SS Antonio Biagio e Cesare Arrigo, Alessandria
  - Ospedale C. e G. Mazzoni UOS Ematologia, Ascoli Piceno
  - Centro di riferimento Oncologico - Oncologia Medica A, Aviano (PN)
  - SOS Ematologia Divisione Medicina Interna Ospedale degli Infermi, Biella
  - Divisione di Ematologia Spedali Civili, Brescia
  - A.O. Universitaria Ospedale Vittorio Emanuele E Ferrarotto Di Catania, Catania
  - AO Santa Croce e Carle, Cuneo
  - A.O. Universitaria Careggi Di Firenze, Florence
  - A.S.L. 9 Opsedali Riuniti del Canavese, Ivrea
  - Area Vasta Romagna e IRST, Meldola (FC)
  - A O Papardo, Messina
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - A.O. Universitaria Policlinico Di Modena, Modena
  - AOU Maggiore della Carità di Novara, Novara
  - IRCCS Istituto Oncologico Veneto -Oncologia 1, Padua
  - Ausl Di Piacenza, Piacenza
  - AO Arcispedale S.Maria Nuova Ematologia, Reggio Emilia
  - AOU La Sapienza, Roma
  - Nuovo Ospedale Civile di Sassuolo - Day Hospital Oncologico, Sassuolo
  - A.O. Universitaria Citta' Della Salute E Della Scienza Di Torino, Torino
  - A.O.U. Citta della Salute e della Scienza di Torino - Ematologia Universitaria, Torino
  - Ematologia - OSPEDALE DI CIRCOLO E FONDAZIONE MACCHI, Varese